CLINICAL TRIAL: NCT03232918
Title: A Randomized Controlled Trial Evaluating the Effect of the Oxytocin Infusion Rate on Fetal Heart Rate Changes and Maternal-Fetal Outcomes During the Initiation of Combined Spinal-Epidural Labor Analgesia
Brief Title: Oxytocin and Fetal Heart Rate Changes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Unyime Ituk (Other)
Responsible Party: Sponsor-Investigator, Unyime Ituk, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201609722
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Fetal Bradycardia Complicating Labor and Delivery; Fetal Bradycardia During Labor; Fetal Heart Rate or Rhythm Abnormality Affecting Fetus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The labor room nurse will be aware of the patient group assignment and will adjust the dose of the drug based on group assignment. The Investigator, Physician Provider and Outcome Assessor will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Dose Oxytocin (No Intervention): Patients randomized to the standard dose oxytocin will have their oxytocin infusion maintained at the standard of care protocol prior to placement of a combined spinal epidural for labor analgesia
- Half Dose Oxytocin (Experimental): Patients randomized to the half dose oxytocin will have their oxytocin infusion reduced by 50 % prior to placement of a combined spinal epidural for labor analgesia.
  Interventions: Drug: Half dose Oxytocin

INTERVENTIONS:
Drug: Half dose Oxytocin — Patients randomized to the half dose oxytocin group will have the oxytocin infusion reduced to 50 % prior to placement of combined spinal epidural for labor analgesia
  Arms: Half Dose Oxytocin

SUMMARY:
The reported risk of nonreassuring fetal heart trace following neuraxial analgesia is 3-23%. This variability may be due to fluid and oxytocin management prior to and during the initiation of neuraxial analgesia. The study hypothesis is that decreasing the oxytocin infusion rate by 50 % prior to initiation of combined spinal epidural analgesia will cause a reduction in the incidence of adverse fetal heart rate changes.

DETAILED DESCRIPTION:
Oxytocin is used in labor and delivery to increase the frequency of contractions and augment uterine contractile strength, thereby establishing a regular pattern of labor. However, the administration of exogenous oxytocin in the presence of an uncoordinated labor pattern confers a risk for an increase in uterine contraction frequency, resulting in inadequate relaxation periods. This leads to an increase in the basal tone of the uterus, which may lead to a tetanic contraction with the risk of decreased uteroplacental blood flow and fetal hypoxemia. Previous studies investigating low- versus high-dose oxytocin for induction or augmentation of labor have had conflicting results on the effect on fetal heart rate abnormalities. One of the limitations of these studies is that the labor analgesia was not standardized. The combination of low-dose combined spinal epidural analgesia and the high/low dose oxytocin have not been evaluated. One of the proposed mechanisms for nonreassuring fetal heart a tracing after initiation of analgesia is that the pain relief from neuraxial analgesia causes a decrease in catecholamine release by the sympathetic nervous system. The subsequent decrease in the circulating epinephrine concentration contributes to an increase in uterine tone, as epinephrine is a potent tocolytic agent. The increased tone, in turn, leads to a decrease in placental blood flow, and eventually fetal bradycardia. The primary outcome of this study is the incidence of non-reassuring fetal heart rate tracings within the first 60 minutes after the placement of combined spinal epidural analgesia

ELIGIBILITY:
Inclusion Criteria:

* Healthy nulliparous or multiparous women at term (37 > weeks' gestation)
* Singleton pregnancy
* Request for neuraxial analgesia
* Oxytocin used for induction of labor or augmentation of labor per institutional protocols

Exclusion Criteria:

* Use of chronic analgesic medications
* Prior administration of systemic opioid labor analgesia
* Non-vertex presentation
* Contraindication to neuraxial analgesia
* Category 3 fetal heart rate tracing prior to the initiation of combined spinal epidural analgesia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 730 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of non-reassuring fetal heart rate tracings | 1.5 hours
  Fetal heart rate tracings will be examined for 30 minutes before and 60 minutes after the initiation of combined spinal epidural analgesia

SECONDARY OUTCOMES:
Effect of oxytocin dose on duration of 1st and 2nd stage of labor | 24 hours
  The effect of the intervention on the duration of labor
Mode of delivery | 24 hours
  The effect of the intervention on the rate of spontaneous vaginal delivery, instrumental vaginal delivery and cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Unyime Ituk, Study Director — University of Iowa
Locations (2):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: CSR
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal

REFERENCES:
- [Background] Mardirosoff C, Dumont L, Boulvain M, Tramer MR. Fetal bradycardia due to intrathecal opioids for labour analgesia: a systematic review. BJOG. 2002 Mar;109(3):274-81. doi: 10.1111/j.1471-0528.2002.01380.x. PMID 11950182
- [Background] Abrao KC, Francisco RPV, Miyadahira S, Cicarelli DD, Zugaib M. Elevation of uterine basal tone and fetal heart rate abnormalities after labor analgesia: a randomized controlled trial. Obstet Gynecol. 2009 Jan;113(1):41-47. doi: 10.1097/AOG.0b013e31818f5eb6. PMID 19104358
- [Background] Clarke VT, Smiley RM, Finster M. Uterine hyperactivity after intrathecal injection of fentanyl for analgesia during labor: a cause of fetal bradycardia? Anesthesiology. 1994 Oct;81(4):1083. doi: 10.1097/00000542-199410000-00041. No abstract available. PMID 7943823
- [Background] Satin AJ, Leveno KJ, Sherman ML, Brewster DS, Cunningham FG. High- versus low-dose oxytocin for labor stimulation. Obstet Gynecol. 1992 Jul;80(1):111-6. PMID 1603479
- [Background] Budden A, Chen LJ, Henry A. High-dose versus low-dose oxytocin infusion regimens for induction of labour at term. Cochrane Database Syst Rev. 2014 Oct 9;2014(10):CD009701. doi: 10.1002/14651858.CD009701.pub2. PMID 25300173